CLINICAL TRIAL: NCT02131818
Title: Necessity of Antibiotics for Prevention of Delivery-associated Infections After Spontaneous Vaginal Delivery at Term
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The enrollment process is too difficult to complete
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SI-OBG-CEU-01-2014
Record Dates: First submitted 2014-04-28; First posted 2014-05-06 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Perineal Wound Infection
Keywords: amoxicillin; postpartum infections; puerperal infection
MeSH Terms: conditions — Puerperal Infection | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amoxicillin (Experimental): The patient will be received amoxicillin 500 mg 2 capsules orally bid pc for 5 days
  Interventions: Drug: Amoxicillin
- Placebo (Placebo Comparator): The patient will be received placebo 2 capsules orally bid pc for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amoxicillin — The patient will be received amoxicillin 500 mg 2 capsules orally bid pc for 5 days
  Other Names: Drug A; Drug B
  Arms: Amoxicillin
Drug: Placebo — The patient will be received placebo 2 capsules orally bid pc for 5 days
  Other Names: Drug A; Drug B
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine amoxicillin is effective in the prevention of wound infection in normal labor.

DETAILED DESCRIPTION:
When the pregnant women is admitted due to first stage of labor , the investigator will inform the patients. If the patients give consent, the patient's data will be collect in case record form. the patients will be swab at posterior fornix and around anus to collect specimen and send to microbiology lab before per vaginal examination. After the patients finish in labor, perineal wound will be swab to collect specimen and send to microbiology lab. Then the patients are randomized in two group, the first one will receive amoxicillin and the second one will receive placebo. During admission the patients will be exam by investigator every day. After the patients are discharge, the follow up will be appoint on 6 weeks later. The infant will be swab at rectum to collect specimen and send to microbiology lab when the patient's discharge day. Every specimen will be culture for bacteria and perform antimicrobial susceptibility test for amoxicillin.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy
* Normal labor

Exclusion Criteria:

* Penicillin allergy
* Previous history antibiotic using within 2 weeks
* Patients cannot take oral medication
* Patients have underlying disease eg. diabetes mellitus, hypertension, HIV infection
* Premature rupture of membranes

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Incidence of perineal wound infection | within 6 weeks after normal labor
  Follow up perineal wound every day during admission and follow up 6 weeks after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Vitaya Titapant, MD, Principal Investigator — Department of Obstetrics & Gynaecology, Faculty of Medicine Siriraj Hospital, Mahidol University, Thailand
Locations (1):
- Faculty of Medicine Siriraj Hoapital Mahidol University, Bangkok, Thailand